CLINICAL TRIAL: NCT01596660
Title: Transversus Abdominis Bilateral Plane Block in Total Laparoscopic Hysterectomy : A Randomized Controlled Trial
Acronym: TAPBLOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Gustavo Adolfo Calle Gomez, Principal investigator, CES University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-JMejia
Record Dates: First submitted 2012-04-30; First posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Block
Keywords: Tap block; laparoscopic hysterectomy; pain
MeSH Terms: conditions — Bites and Stings; Pain | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaina (Experimental): 20 cc of bupivacaine 0.5% in 20 cc de saline solution and it is infiltrated 20 cc each side.
  Interventions: Drug: Bupivacaina 0.5%
- saline solution (Placebo Comparator): 20 cc of saline solution 0.9% to infiltrate each side.
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: Bupivacaina 0.5% — Bupivacaina 0.5% 20cc
  Other Names: Bupivacaine
  Arms: Bupivacaina
Drug: placebo comparator — 20 cc of saline solution 0.9%, to infiltrate each side.
  Other Names: Saline solution
  Arms: saline solution

SUMMARY:
The ambulatory management after laparoscopic hysterectomy is a reality in our service, where 90% of hysterectomies are laparoscopically done and 80% of these are managed on an ambulatory basis with shorter hospital stay ;less than 12 hours. (OALOS 9.41 + / - (1.79) range from 5 to 12 hours and POLE 5.38 + / - (1.8) range from 2 to 9 hours)

So far the immediate analgesic management has been made systemically, and the satisfaction reported by patients was high, even though some patients require longer stay in recovery and need higher doses of analgesics before their discharge criteria, allowing an optimal ambulatory management.

There are several treatment options that theoretically could be used but the results have been variable and have failed to demonstrate the expected benefit.

The Transversus Abdominis Plane Block consists in the deposition of local anesthetic in the plane between the internal oblique and transverse abdominal, looking to infiltrate the spinal nerves at this level, so the innervation to the skin, muscles and the parietal peritoneum will be interrupted. The TAP Block was first described in 2001 , based on anatomy marks techniques of the peripheral nerves and was developed and evaluated later by McDonnell et al.

DETAILED DESCRIPTION:
The blockage in the abdominal transverse plane (TAP Block) with local anesthetic has demonstrated efficacy and safety in patients with various types of abdominal surgery by laparotomy as both laparoscopically.

The blockage in the abdominal transverse plane is a single entry in the triangle of Petit, to access a greater number of nerves that allow a wider spread of analgesia. The innervation of the anterolateral abdominal wall is given by the anterior branches of spinal nerves T7 to L1 (these include the intercostal nerves T7 at 11, the nerve subcostal nerve T12 and ilio hypogastric and ilio inguinal L1

The anterior divisions of the nerves T7 to T11 continues from the intercostal space and enter the abdominal wall between the internal oblique and transversus abdominis, reaching the rectus abdominis, which pierce and innervate the skin of the anterior abdominal region. In its course also innervate the external oblique muscle via the lateral cutaneous branch is divided into anterior and posterior innervating the external oblique and dorsal latium

The anterior branch of T12 is connected to the ilio hypogastric nerve and gives branch to the piriformis muscle, the lateral cutaneous branch pierces the internal and external oblique muscles and descends over the iliac crest innervate the anterior part of the buttocks.

The ilio hypogastric nerve,L1, is divided between the internal oblique and transversus abdominis near the iliac crest in two anterior and lateral cutaneous branches, the first innervate the skin of the buttocks and the second the hypogastric region.

The ilio inguinal nerve communicates with the ilio hypogastric nerve between the internal oblique and transversus abdominis, near the anterior iliac crest and innervates the anterior and medial thigh and part of the skin covering the genitals.

The aim of the nerve block is to deposit local anesthetic in the plane between the internal oblique and transverse abdominal looking to infiltrate the spinal nerves at this level, so the skin innervation on muscle and parietal peritoneum will interrupted. Obviously if the surgery goes through the peritoneal cavity, visceral pain will not be interrupted.

This block is indicated in any lower abdominal surgery and has been used effectively in laparoscopic surgery, so far no work described in LH, this block allows analgesia from T7 to L1 even with minimal side effects, low cost, without altering surgical time, and low risk. Among the complications described above, a puncture of the liver in a patient with liver elongated and some small punctures without serious consequences.

The ambulatory management could be more efficient with the use of blockage in the abdominal transverse plane (TAP Block) with local anesthetic. In order to study the benefits that the TAP Block could offer to our patients, we suggest a randomized controlled trial comparing the blockage in the abdominal transverse plane with placebo.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for laparoscopic hysterectomy for benign causes.
* ASA 1 and 2
* Patients without contraindications to the administration of local anesthetics
* Patients without contraindications to NSAIDs or acetaminophen.
* Patients with no simultaneous intervention (only laparoscopic hysterectomy)
* Patients living in the metropolitan area, with telephone line, can be contacted by telephone in the first 72 hours by calling 24, 48 and 72 hours, conducted by researchers at the number previously reported by the patient.
* An adequate level of understanding, ie patients who are able to communicate by telephone and understand a numerical scale.
* Who agree to participate in the work.

Exclusion Criteria:

* Patients who should undergo a change in the standard anesthetic technique.
* Patients who are hospitalized after total laparoscopic hysterectomy.
* Patients with a body mass index above 30.
* Laparoscopic hysterectomy with a longer duration to 120 minutes.
* Patients who do not they can be reached by phone at pre-set times.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hours
  The instrument used to assess pain intensity is a straight line marked with numbers 1 to 10, with 1 meaning absence of pain and 10 the worst pain imaginable. The patient marks a point on the line that matches the pain she feels.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A Calle, MD, Study Director — CES University
Locations (1):
- Universidad CES, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Lenz H, Sandvik L, Qvigstad E, Bjerkelund CE, Raeder J. A comparison of intravenous oxycodone and intravenous morphine in patient-controlled postoperative analgesia after laparoscopic hysterectomy. Anesth Analg. 2009 Oct;109(4):1279-83. doi: 10.1213/ane.0b013e3181b0f0bb. PMID 19762758
- [Background] Scharine JD. Bilateral transversus abdominis plane nerve blocks for analgesia following cesarean delivery: report of 2 cases. AANA J. 2009 Apr;77(2):98-102. PMID 19388503
- [Background] Malhotra N, Chanana C, Roy KK, Kumar S, Rewari V, Sharma JB. To compare the efficacy of two doses of intraperitoneal bupivacaine for pain relief after operative laparoscopy in gynecology. Arch Gynecol Obstet. 2007 Oct;276(4):323-6. doi: 10.1007/s00404-007-0337-1. Epub 2007 Jul 25. PMID 17653742
- [Background] de Lapasse C, Rabischong B, Bolandard F, Canis M, Botchorischvili R, Jardon K, Mage G. Total laparoscopic hysterectomy and early discharge: satisfaction and feasibility study. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):20-5. doi: 10.1016/j.jmig.2007.08.608. PMID 18262139
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] Jankovic ZB, Pollard SG, Nachiappan MM. Continuous transversus abdominis plane block for renal transplant recipients. Anesth Analg. 2009 Nov;109(5):1710-1. doi: 10.1213/ANE.0b013e3181ba75d1. No abstract available. PMID 19843821
- [Background] Fredrickson MJ, Seal P. Ultrasound-guided transversus abdominis plane block for neonatal abdominal surgery. Anaesth Intensive Care. 2009 May;37(3):469-72. doi: 10.1177/0310057X0903700303. PMID 19499870
- [Background] Niraj G, Kelkar A, Fox AJ. Application of the transversus abdominis plane block in the intensive care unit. Anaesth Intensive Care. 2009 Jul;37(4):650-2. doi: 10.1177/0310057X0903700420. PMID 19681428
- [Result] Preliminary experience with transversus abdominis plane block for postoperative pain relief in infants and children